CLINICAL TRIAL: NCT00823966
Title: Drug Use Investigation For Rescriptor (Regulatory Post Marketing Commitment Plan)
Brief Title: Safety And Efficacy Of Rescriptor In Patients For Human Immunodeficiency Virus (HIV) Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A4351010
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-06

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Delavirdine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Delavirdine Mesilate: Patients administered.
  Interventions: Drug: Rescriptor

INTERVENTIONS:
Drug: Rescriptor — RESCRIPTOR® TABLETS 200mg, depending on the Investigator prescription. Frequency and duration are according to Package Insert as follows. "The usual adult dose is 400mg of Delavirdine Mesilate administered orally 3 times daily.This drug must always be administered in combination with other anti-HIV drugs."
  Other Names: Rescripter

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the Local Product Document (LPD) (unlisted adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Rescriptor® should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

Patients need to be administered Rescriptor® in order to be enrolled in the surveillance.

Exclusion Criteria:

Patients not administered Rescriptor®.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A4351010 prescribes the Delavirdine Mesilate(Rescriptor).
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2003-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4351010&StudyName=Safety%20And%20Efficacy%20Of%20Rescriptor%20In%20Patients%20For%20HIV%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 08 December 2003 to 31 March 2009, a total of two centers in Japan
Groups:
- Delavirdine Mesilate: RESCRIPTOR® TABLETS 200mg, depending on the Investigator prescription. Frequency and duration are according to Package Insert as follows. "The usual adult dose is 400mg of Delavirdine Mesilate administered orally 3 times daily.This drug must always be administered in combination with other anti-human immunodeficiency virus (HIV) drugs."
Period: Overall Study
Arm/Group | Delavirdine Mesilate
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Delavirdine Mesilate
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  Japan | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Unlisted Adverse Drug Reaction.
Description: Adverse drug reaction that is not listed in the Japanese Package Insert(Same as Local product Document).
Time Frame: One Year
Population: The safety analysis population included enrolled subjects who had received at least 1 confirmed, administration of delavirdine mesylate.
Measure: Number; unit: participants
Arm/Group | Delavirdine Mesilate
Number analyzed (Participants) | 3
participants | 0

2. Primary Outcome: Number of Participants Who Improved in Number of HIV- Ribonucleic Acid (RNA) Copies, Cluster of Differentiation 4(CD4) Count, and Not Progress in HIV Classification: Centers for Disease Control and Prevention Clinical Category (CDC Category).
Description: Improvement of number of HIV-RNA copies; Improvement is measured by general evaluation of decrease in HIV-RNA copies.
  Improvement of CD4 counts; Improvement is measured by general evaluation of increase in CD4 counts.
  Not progress in HIV classification (severity of CDC category); Subjects were classified based on the severity of CDC category as mild (Category A), moderate (Category B), and severe (Category C). No change categories from Category A to Category B / Category C, or from Category B to Category C in CDC category.
Time Frame: One year
Population: The efficacy analysis population included all subjects from the safety analysis population in whom the efficacy of this drug could be evaluated.
Measure: Number; unit: participants
Arm/Group | Delavirdine Mesilate
Number analyzed (Participants) | 3
participants
  Number of HIV-RNA | 3
  CD4 | 2
  CDC category | 3

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Delavirdine Mesilate
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delavirdine Mesilate (N=3)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delavirdine Mesilate (N=3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There is not enough data to analyze on the efficacy and safety of delavirdine mesylate in the 3 subjects with HIV infection assessed during this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes